CLINICAL TRIAL: NCT02878525
Title: Study the Effectiveness and Safety of Laparoscopic Internal Gastric Banding, New Simple and Costless Weight Loss Procedure, in Comparison to Laparoscopic Sleeve Gastrectomy
Brief Title: Laparoscopic Internal Gastric Banding, New Simple and Costless Weight Loss Procedure
Acronym: LIGB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Mstafa Hassan Sewefy, MD, Lecturer & consultant of general surgery, Department of surgery, Minia university hospital, Egypt, Minia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: fac.med.018
Record Dates: First submitted 2016-08-21; First posted 2016-08-25 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic internal gastric banding (Experimental): Laparoscopic internal gastric banding
  Interventions: Procedure: Laparoscopic internal gastric banding
- Laparoscopic sleeve gastrectomy (Active Comparator): Laparoscopic sleeve gastrectomy
  Interventions: Procedure: laparoscopic sleeve gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic internal gastric banding — Laparoscopic internal gastric banding
  Arms: Laparoscopic internal gastric banding
Procedure: laparoscopic sleeve gastrectomy — laparoscopic sleeve gastrectomy
  Arms: Laparoscopic sleeve gastrectomy

SUMMARY:
The purpose of this study is to study the effectiveness of laparoscopic internal gastric banding as a treatment for morbid obesity in comparison to laparoscopic sleeve gastrectomy

DETAILED DESCRIPTION:
In this study 190 morbidly obese patients will be included and will randomly assign into 2 groups, group 1 will be operated by laparoscopic internal gastric banding and group 2 by laparoscopic sleeve gastrectomy, the patients will be followed up for 1 year to evaluate the effectiveness and drawbacks of laparoscopic internal gastric banding in comparison to laparoscopic sleeve gastrectomy, the investigators preparing to submit our study protocol to our institution ethical committee for approval to start the study

ELIGIBILITY:
Inclusion Criteria:

* BMI more than 40 with or without co-morbidity or more than 35 with co-morbidity
* Approval to share in the study
* Patients fit for laparoscopic surgery

Exclusion Criteria:

* Patient age less than 18 or more than 50 years old
* Refusal to share in the study
* Unfit for surgery
* patients with gastroesophageal reflux disease clinically or by investigation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2016-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
safety of the technique | 4 weeks
  the incidence of introperative and early postoperative complications

SECONDARY OUTCOMES:
operative time | 12 hours
  the operative time from skin to skin
Hospital stay | 30 days
  Time of hospital stay
total cost | 16 weeks
  the total cost of the technique by US dollar and its early complications
Metabolic effect | 6-12 months
  Effect of the procedure on blood sugar, serum lipid and hypertension

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of medicine, Minya
  - Minia university hospital, Minya

IPD SHARING:
Plan to Share IPD: Undecided